CLINICAL TRIAL: NCT06313749
Title: An Observer-Masked, Single-Arm, Multicenter Study to Evaluate the Safety and Effectiveness of Minimally Invasive Micro Sclerostomy (MIMS®) to Reduce Intraocular Pressure in Open-Angle Glaucoma Which is Not Controlled Despite Polypharmacy
Brief Title: Safety and Effectiveness of Minimally Invasive Micro Sclerostomy (MIMS®) to Reduce Intraocular Pressure in Open-Angle Glaucoma Which is Not Controlled Despite Polypharmacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMS-US-1
Record Dates: First submitted 2024-03-02; First posted 2024-03-15 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Primary Open Angle Glaucoma; Open Angle Glaucoma
Keywords: Open Angle Glaucoma; Polypharmacy; Intraocular Pressure; MIMS; Minimally Invasive Glaucoma Surgery; MIGS; MTMT
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Masking Description: This clinical study is observer masked only when measuring intraocular pressure (using Goldmann Applanation Tonometry). Intraocular pressure measurements will be determined using the 2-person method to reduce bias. Observer 1 (masked to real time reading) will look through the slit lamp and turn the Goldmann Tonometer dial, and Observer 2 will read and record the intraocular pressure readings. Observer 1 will be unable to see the readings with the use of a masking card.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MIMS® Device/Procedure Arm (Experimental): Arm which includes subjects undergoing the MIMS® surgical procedure using the proprietary MIMS® device developed by Sanoculis Ltd.
  Interventions: Device: Minimally Invasive Micro Sclerostomy Device

INTERVENTIONS:
Device: Minimally Invasive Micro Sclerostomy Device — During this clinical trial, the Minimally Invasive Micro Sclerostomy (MIMS®) procedure will be performed by investigators using the proprietary MIMS® device developed by Sanoculis Ltd.
  Other Names: MIMS® Device

SUMMARY:
The goal of this clinical trial is to show non-inferiority of the MIMS® device/procedure with Mitomycin-C, in terms of its surgical success rate, compared to trabeculectomy with Mitomycin-C in subjects diagnosed with primary open angle glaucoma, whose intraocular pressure is not controlled despite polypharmacy.

Eligible screened participants will undergo the MIMS® procedure and will be followed for a period of 12 months in this single-arm study. Investigators will compare the results of this study to the surgical success rate of traditional trabeculectomy with Mitomycin-C.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 40 years to ≤ 85 years old
2. Inadequately controlled primary open angle glaucoma with screening mean diurnal IOP of ≥ 21 mmHg and ≤ 40 mmHg despite polypharmacy
3. Primary open angle glaucoma diagnosis based on:

   1. Visual field mean deviation of -3dB or worse and
   2. Glaucomatous optic nerve damage as evidenced by optic disc or retinal nerve fiber layer structural abnormalities documented on slit lamp stereo biomicroscopy or in stereo disc photos
4. Presence of healthy, free, and mobile conjunctiva in the target quadrant
5. Prior ab interno conjunctival-sparing glaucoma procedures were conducted more than 6 months prior to enrollment (e.g., iStent, Trabectome, gonioscopy-assisted transluminal trabeculectomy [GATT])
6. Subject is able and willing to attend all scheduled follow-up exams
7. Subject understands and signs the informed consent

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate of the MIMS® device/procedure at 12 months after surgery | 12 months
  Definition of Surgical Success: the subject's eye, after having the MIMS® procedure:
  1. Achieved 20% or more reduction in average diurnal IOP from baseline at 12 months after surgery; AND
  2. Using the same number or fewer topical IOP lowering medications

SECONDARY OUTCOMES:
Exploratory Effectiveness Endpoint 1 | 12 months
  Change in IOP (mmHg) from baseline to 12 months follow-up
Exploratory Effectiveness Endpoint 2 | 12 months
  Change in IOP (% change) from baseline to 12 months follow-up
Exploratory Effectiveness Endpoint 3 | 12 months
  Change in the number of IOP lowering topical medications from screening to 12 months follow-up
Exploratory Effectiveness Endpoint 4 | 12 months
  Change in number (% change) of IOP lowering topical medications from screening to 12 months follow-up
Safety Outcome 1 | 12 months
  Incidence of ocular adverse events in the study eye (overall and related to MIMS® device/procedure) throughout the follow-up period
Safety Outcome 2 | 12 months
  Biomicroscopic slit lamp and ophthalmoscopy findings
Safety Outcome 3 | 12 months
  Preservation of Best-Corrected Visual Acuity (BCVA)

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Associates of Texas, Dallas, Texas, United States